CLINICAL TRIAL: NCT06295848
Title: The Effects of 6-week Cardiac Rehabilitation Programme on Cardiovascular Disease Risk, Systolic and Diastolic Blood Pressure and Disease Activity in Hypertensive Rheumatoid Arthritis Patients : A Randomised Controlled Trial
Brief Title: The Effects of Cardiac Rehabilitation Programme in Hypertensive Rheumatoid Arthritis Patients
Acronym: CARDIRA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kayseri City Hospital (Other Government)
Responsible Party: Principal Investigator, Havva Talay Çalış, Professor Doctor, Kayseri City Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KayseriCH005
Record Dates: First submitted 2023-09-01; First posted 2024-03-06 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: Cardiac Rehabilitation; Rheumatoid Arthritis; Hypertension
MeSH Terms: conditions — Arthritis, Rheumatoid; Hypertension | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cardiac Rehabilitation (Experimental): The CR group will receive training for CVD and HT once a week, along with a rehabilitation program consisting of aerobic, resistance, flexibility and stretching exercises 3 days a week for 6 weeks.
  Interventions: Behavioral: Exercise
- Control (No Intervention): Control group will receive treatment for their RA that is considered standard of care treatment (e.g. pharmacotherapy), but will not be participated in the CR program.

INTERVENTIONS:
Behavioral: Exercise — An individual program will be organized for each patient according to the exercise test result. Since the patients have both arthritis and HTN, aerobic exercises will be given at moderate intensity (40-60% VO2 reserve) according to ACMS recommendations. Xrcise Runner Med treadmill and Xrcise Care 2.5.8.3 software will be used for aerobic exercises. Resistant exercises will be given under the supervision of a physiotherapist, calculating 1 repetitation maximum (1-RM) in the main muscle groups.Patients will perform isotonic exercises with 3 sets of 15 repetitions with a resistance of 60% of 1-RM. The education sessions will be conducted by a multidisciplinary team of health professionals (nurse, physiotherapist and dietician) under the leadership of a clinician experienced in CR. Education topics will consist of 60-minute sessions covering heart-healthy eating, setting health-related goal, exercise, diet, healthy weight loss, smoking cessation, and stress/coping.
  Arms: Cardiac Rehabilitation

SUMMARY:
The aim of this study is to investigate the beneficial impacts of the 6-week standardized CR program applied to hypertensive RA patients whose disease activity is under control with regular pharmacological treatment.

Subjects will be randomly assigned to one of two groups: 1.) standard of care (SOC) treatment or 2.) SOC plus a 6 week CR program.

DETAILED DESCRIPTION:
Rheumatoid arthritis (RA) is a chronic systemic auto-immune disease characterized by inflammation and structural damage in synovial joints, but also has extra-articular involvements such as the cardiovascular system. RA patients have higher mortality rates than the general population, and approximately half of premature deaths are due to cardiovascular comorbidities. Traditional risk factors, especially hypertension (HTN), play a key role in the development of cardiovascular diseases (CVD).

In chronic inflammatory diseases such as RA, autoimmunity is a cause of HTN as well as a result of physical damage to the vascular wall. Mild blood pressure elevation caused by specific HTN triggers such as salt retention, angiotensin-II or genetic susceptibility leads to neoantigen release through tissue damage. These neoantigens are recognized by antigen-presenting cells and lead to the differentiation of CD4+ naïve-T lymphocytes into Th1 and Th17 cells. IL-17 and IFN-γ expression causes local inflammation in the vascular wall, endothelial dysfunction, and arterial stiffness. Thus, HTN causes an increase in CVD risk through a common pathogenesis mechanism with RA.

European League Against Rheumatism (EULAR) recommendations emphasize that rheumatologists should be responsible for CVD risk management in RA. However, both RA and HTN treatment is generally administered pharmacologically without focusing on CVD risk. Patients may be recommended regular exercise and lifestyle changes according to EULAR recommendation guide for CVD risk management. One possible intervention that could be used to decrease CVD risk caused by both diseases is cardiac rehabilitation (CR) program in which regular exercise is one of the main components. But RA patients, especially those with cardiovascular comorbidities, are rarely referred to the CR program.

This study will help to clarify the effects of the CR program added to the pharmacological treatment of these patients on cardiovascular mortality risk (Framingham risk score and QRISK-3 score), blood pressure (24-Hour holter monitoring), disease activity (DAS28-CRP), aerobic capacity (VO2max), quality of life (36-Item Short Form Survey) and psychological state (Beck depression inventory).

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with RA according to ACR/EULAR 2010 criteria
2. Taking regular treatment for at least 1 month according to ACR/EULAR guidelines
3. Patients diagnosed with HT according to the 2018 European Society of Hypertension and European Society of Cardiology (ESH/ESC) guideline

Exclusion Criteria:

1. Refusing to participate in the program
2. Severe mental disorder
3. Neurological disease or deformity in the lower extremity that would prevent the patient from using the treadmill.
4. High-risk unstable angina and all acute cardiac diseases (acute myocardial infarction, acute endocarditis, myocarditis or pericarditis)
5. Uncontrolled HT, Diabetes, cardiac arrhythmia and heart failure
6. Symptomatic severe aortic stenosis
7. Acute pulmonary embolism or pulmonary infarction and severe pulmonary hypertension

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-12-15 (Actual); Primary Completion 2024-04-15 (Estimated); Study Completion 2024-06-15 (Estimated)

PRIMARY OUTCOMES:
Framingham Risk Score(FRS) | 0-week, 6-week,12-week,24-week
  It is a common tool used to assess a patient's risk level of cardiovascular disease over the next 10 years. There are six coronary risk factors in the FRS calculation, including age, gender, total cholesterol, HDL cholesterol, smoking and systolic blood pressure. 10-year cardiovascular risk score can be derived as a percentage. Higher values indicate a worse, lower values indicate a better outcome.
QRISK-3 Risk Score | 0-week, 6-week,12-week,24-week
  It predicts a patient's risk of developing cardiovascular disease in the next 10 years. It includes many of the traditional risk factors featured in Framingham (such as age, gender, cholesterol/HDL ratio, blood pressure, diabetes and smoking status), but also includes important additional risk factors. 10-year cardiovascular risk score can be derived as a percentage. Higher values indicate a worse, lower values indicate a better outcome.
24-Hour Ambulatory Blood Pressure | 0-week, 6-week,12-week,24-week
  It is the gold standard for hypertension diagnosis and 24-hour blood pressure evaluation.
DAS28 | 0-week, 6-week,12-week,24-week
  Rheumatoid arthritis severity will be determined using DAS28 score. The DAS28 score ranges score between 0 and 10, a larger number indicating more active disease. When using the score to assess response to treatment, a DAS-28 score reduction by 0.6 represents a moderate improvement, while a reduction more than 1.2 represents a major improvement. The score <2.6 suggests disease remission.
Maximal oxygen consumption (VO2max) | 0-week, 6-week,12-week,24-week
  VO2 max is the number of milliliters of oxygen used per kilogram of body weight in one minute (ml/kg/min). VO2 max is an objective measurement of cardiorespiratory capacity. Higher values indicate a worse, lower values indicate a better outcome.

SECONDARY OUTCOMES:
The Six-Minute Walk Test (6MWT) | 0-week, 6-week,12-week,24-week
  The Six-Minute Walk Test is a submaximal field test used to monitor exercise capacity and treatment effectiveness in cardiac rehabilitation.
The 36-Item Short Form Survey (SF-36) | 0-week, 6-week,12-week,24-week
  Quality of life will be assessed using the short form of the 36-Item short form survey (SF-36). The SF-36 covers eight health concepts: physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, emotional well-being, social functioning, energy/fatigue, and general health perceptions. Scores for each domain range from 0 to 100, with a higher score defining a more favorable health state.
International Physical Activity Questionnaire (IPAQ) - Short Form | 0-week, 6-week,12-week,24-week
  The IPAQ short form encompasses questions regarding time spent on walking, moderate-intensity, and high-intensity physical activities besides sitting. The IPAQ scoring protocol assigns the following MET values to walking, moderate, and vigorous intensity activity: 3.3 METs, 4.0 METs, and 8.0 METs, respectively. Total physical activity can be computed as the sum of walking + moderate intensity + high intensity MET-min/week scores. Higher values indicate a worse, lower values indicate a better outcome. There are three levels of physical activity suggested for classifying patients based on total weekly MET score: low, moderate and high. The "minutes" of sitting reported by the IPAQ are asessed independtly and reflect sedentary behaviour measurements.
Beck Depression Inventory (BDI) | 0-week, 6-week,12-week,24-week
  The Beck Depression Inventory (BDI) is a 21-item, self-report rating inventory that measures characteristic attitudes and symptoms of depression. The minimum score is 0 and maximum score is 63. Higher scores indicate greater symptom severity.

CONTACTS AND LOCATIONS:
Overall Officials: Serap TOMRUK SÜTBEYAZ, PROFESSOR, Study Director — KAYSERİ CITY HOSPITAL; Abdurrahman KUTLUCA, MD, Principal Investigator — Health Sciences University, Kayseri Medical Faculty
Locations (1):
- Health Sciences University, Kayseri Medicine Faculty, Kayseri, Kocasinan, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chauhan K, Jandu JS, Brent LH, Al-Dhahir MA. Rheumatoid Arthritis. 2023 May 25. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK441999/ PMID 28723028
- [Background] Gibofsky A. Epidemiology, pathophysiology, and diagnosis of rheumatoid arthritis: A Synopsis. Am J Manag Care. 2014 May;20(7 Suppl):S128-35. PMID 25180621
- [Background] Almutairi K, Nossent J, Preen D, Keen H, Inderjeeth C. The global prevalence of rheumatoid arthritis: a meta-analysis based on a systematic review. Rheumatol Int. 2021 May;41(5):863-877. doi: 10.1007/s00296-020-04731-0. Epub 2020 Nov 11. PMID 33175207
- [Background] Avina-Zubieta JA, Choi HK, Sadatsafavi M, Etminan M, Esdaile JM, Lacaille D. Risk of cardiovascular mortality in patients with rheumatoid arthritis: a meta-analysis of observational studies. Arthritis Rheum. 2008 Dec 15;59(12):1690-7. doi: 10.1002/art.24092. PMID 19035419
- [Background] Sokka T, Abelson B, Pincus T. Mortality in rheumatoid arthritis: 2008 update. Clin Exp Rheumatol. 2008 Sep-Oct;26(5 Suppl 51):S35-61. PMID 19026144
- [Background] Hadwen B, Stranges S, Barra L. Risk factors for hypertension in rheumatoid arthritis patients-A systematic review. Autoimmun Rev. 2021 Apr;20(4):102786. doi: 10.1016/j.autrev.2021.102786. Epub 2021 Feb 18. PMID 33609791
- [Background] Anyfanti P, Gkaliagkousi E, Triantafyllou A, Koletsos N, Gavriilaki E, Galanopoulou V, Aslanidis S, Douma S. Hypertension in rheumatic diseases: prevalence, awareness, treatment, and control rates according to current hypertension guidelines. J Hum Hypertens. 2021 May;35(5):419-427. doi: 10.1038/s41371-020-0348-y. Epub 2020 May 7. PMID 32382031
- [Background] Jagpal A, Navarro-Millan I. Cardiovascular co-morbidity in patients with rheumatoid arthritis: a narrative review of risk factors, cardiovascular risk assessment and treatment. BMC Rheumatol. 2018 Apr 11;2:10. doi: 10.1186/s41927-018-0014-y. eCollection 2018. PMID 30886961
- [Background] Panoulas VF, Metsios GS, Pace AV, John H, Treharne GJ, Banks MJ, Kitas GD. Hypertension in rheumatoid arthritis. Rheumatology (Oxford). 2008 Sep;47(9):1286-98. doi: 10.1093/rheumatology/ken159. Epub 2008 May 8. PMID 18467370
- [Background] Sahin AA, Ozben B, Sunbul M, Yagci I, Sayar N, Cincin A, Gurel E, Tigen K, Basaran Y. The effect of cardiac rehabilitation on blood pressure, and on left atrial and ventricular functions in hypertensive patients. J Clin Ultrasound. 2020 Dec 1:e22956. doi: 10.1002/jcu.22956. Online ahead of print. PMID 33289108
- [Background] Whelton SP, Chin A, Xin X, He J. Effect of aerobic exercise on blood pressure: a meta-analysis of randomized, controlled trials. Ann Intern Med. 2002 Apr 2;136(7):493-503. doi: 10.7326/0003-4819-136-7-200204020-00006. PMID 11926784
- [Background] Agca R, Heslinga SC, Rollefstad S, Heslinga M, McInnes IB, Peters MJ, Kvien TK, Dougados M, Radner H, Atzeni F, Primdahl J, Sodergren A, Wallberg Jonsson S, van Rompay J, Zabalan C, Pedersen TR, Jacobsson L, de Vlam K, Gonzalez-Gay MA, Semb AG, Kitas GD, Smulders YM, Szekanecz Z, Sattar N, Symmons DP, Nurmohamed MT. EULAR recommendations for cardiovascular disease risk management in patients with rheumatoid arthritis and other forms of inflammatory joint disorders: 2015/2016 update. Ann Rheum Dis. 2017 Jan;76(1):17-28. doi: 10.1136/annrheumdis-2016-209775. Epub 2016 Oct 3. PMID 27697765
- [Background] Metsios GS, Stavropoulos-Kalinoglou A, Veldhuijzen van Zanten JJ, Treharne GJ, Panoulas VF, Douglas KM, Koutedakis Y, Kitas GD. Rheumatoid arthritis, cardiovascular disease and physical exercise: a systematic review. Rheumatology (Oxford). 2008 Mar;47(3):239-48. doi: 10.1093/rheumatology/kem260. Epub 2007 Nov 28. PMID 18045810
- [Background] Peynirci Cersit H, Yagci I, Cersit S. The improvement in aerobic capacity, disease activity, and function in patients with rheumatoid arthritis following cardiac rehabilitation program: A single-center, controlled study. Turk J Phys Med Rehabil. 2019 Apr 26;66(2):121-133. doi: 10.5606/tftrd.2020.3250. eCollection 2020 Jun. PMID 32760888
- [Background] Tessler J, Ahmed I, Bordoni B. Cardiac Rehabilitation. 2025 Mar 28. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK537196/ PMID 30725881
- [Background] Balady GJ, Ades PA, Comoss P, Limacher M, Pina IL, Southard D, Williams MA, Bazzarre T. Core components of cardiac rehabilitation/secondary prevention programs: A statement for healthcare professionals from the American Heart Association and the American Association of Cardiovascular and Pulmonary Rehabilitation Writing Group. Circulation. 2000 Aug 29;102(9):1069-73. doi: 10.1161/01.cir.102.9.1069. No abstract available. PMID 10961975